CLINICAL TRIAL: NCT01906333
Title: Effects of Acute Elevation of Circulating Fatty Acids on Skeletal Muscle Lipid Accumulation and Metabolism in Healthy Lean Young Men
Brief Title: Elevated FFA and Skeletal Muscle Lipid Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lena Bilet, PhD student, Maastricht University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NL43302.068.13/METC 13-3-003
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes; Exercise Physiology
Keywords: Exercise; Ectopic fat accumulation
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Exercise; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise & Glucose (Experimental): 2 hour exercise while getting glucose-supplementation
  Interventions: Other: Exercise; Other: Glucose
- Exercise & Fasted (Experimental): 2 hour exercise while staying fasted
  Interventions: Other: Exercise; Other: Fasted

INTERVENTIONS:
Other: Exercise
Other: Glucose
  Arms: Exercise & Glucose
Other: Fasted
  Arms: Exercise & Fasted

SUMMARY:
There is increasing evidence that skeletal muscle lipid content (IntraMyoCellular Lipid, IMCL) markedly increases the risk of metabolic complications, including insulin resistance and cardiovascular events. The investigator hypothesizes that skeletal muscle is passively taking up FFAs when the availability is high, thereby leading to an increased storage. To test this hypothesis, the investigator wants to manipulate FFA levels, by means of exercise, and monitor intramuscular lipid content.

Therefore the objective is to examine the effect of an exercise-induced elevation of FFA on skeletal muscle lipid content in healthy lean men. To this end, skeletal muscle lipid content will be investigated at baseline and after an exercise protocol and again after a four-hour recovery period from exercise, once in a condition with high FFA concentration, once with low FFA concentration. To achieve high- versus low FFA concentrations, an exercise protocol was chosen and participants had to perform this protocol once with a glucose supplementation and once without.

Skeletal muscle lipid content will be determined before, directly after exercise and 4 h post exercise (from muscle biopsies) with or without glucose supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18-30 years
* Lean, BMI 18-25 kg/m2
* Healthy
* Stable dietary habits
* No medication use

Exclusion Criteria:

* Female sex
* Engagement in programmed exercise > 2 hours total per week
* Cardiac problems, such as angina pectoris, cardiac infarction and arrhythmias
* First degree relatives with type 2 diabetes mellitus
* Any medical condition requiring treatment and/or medication use
* Unstable body weight (weight gain or loss > 3 kg in the past three months)
* Participation in other biomedical study within 1 month prior to the screening visit
* Subjetcs, who do not want to be informed about unexpected medical findings, or do not wish that their treating physician is informed, cannot participate in the study

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in IntraMyoCellularLipid (IMCL)content | Baseline, directly postexercise and 4 hours post-exercise
  A muscle biopsy will be withdrawn before, after 2 hours of exercise and again 4 hours post-exercise for later analysis of IMCL.

SECONDARY OUTCOMES:
Change in substrate metabolism | Measured several time points during the test day
  Substrate metabolism will be measured for 15 min every 30 min of exercise and 20 min every hour of recovery for later analysis of fat- and glucose oxidation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Biology, Maastricht University Medical Center (MUMC), Maastricht, Netherlands